CLINICAL TRIAL: NCT06396767
Title: Diaphragmatic Inspiratory Amplitude Measured by Ultrasonography as a Prognosticator for Postoperative Pulmonary Complications After Cardiac Surgery: a Prospective Observational Cohort Study
Brief Title: Diaphragmatic Inspiratory Amplitude as a Prognosticator for Postoperative Pulmonary Complications After Cardiac Surgery
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Raffael Zamper, Anesthesiologist, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: DIA for POPC
Record Dates: First submitted 2024-04-30; First posted 2024-05-02 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Pulmonary Complications; Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DIA measured via Ultrasonography: Ultrasonographic measurements will be done preoperatively a day before surgery (T0) and on Postoperative day 1(T1) in Cardiac Surgery Recovery Unit (CSRU). Measurements will be done on both right and left sides during Quiet (Q) and Deep (D) breathing in semi- recumbent posture (30-450 recline of the bed).
  Three measurements will be taken during both quiet and deep breathing and an average value will be derived (Qavg and Davg). this will be done for both right and left hemidiaphragms (both pre-surgery and post-surgery). So, for each patient a total of 8 diaphragmatic measurements will be obtained (4 in the pre-surgery period and another 4 in post-surgery period). Measurement technique and definition of Diaphragmatic Inspiratory Amplitude:
  All examinations will be performed by Sonosite SII ultrasound machine (FUJIFILM Sonosite Inc, Bothell, WA, USA) using a 3.5- to5 MHz phased array probe or a 3-12 MHz linear probe.
  Interventions: Diagnostic Test: DIA measured via Ultrasonography

INTERVENTIONS:
Diagnostic Test: DIA measured via Ultrasonography — Ultrasound will be used to measure Diaphragmatic Inspiratory Amplitude (DIA) of patients before and after elective cardiac surgery to determine if there is a correlation between changes in DIA and postoperative pulmonary complications.

SUMMARY:
Cardiac surgery is a critical intervention for a variety of cardiovascular conditions, yet it can frequently results in a spectrum of postoperative complications. Amongst various morbidities, Post-Operative Pulmonary Complications (POPCs) represent a significant clinical challenge leading to adverse outcomes like increased morbidity, mortality, and raised healthcare expenditures. The diaphragm, as the principal respiratory muscle, plays a pivotal role in maintaining pulmonary function. Diaphragmatic dysfunction (DD) in the perioperative period of Cardiac surgery has an incidence of up to 20%. Understanding the impact of DD on postoperative pulmonary function is imperative for optimizing patient care and clinical outcomes. Its occurrence has been linked to a spectrum of respiratory complications, ranging from pneumonia to difficulty in weaning from mechanical ventilation. In recent years, the advent of point-of-care ultrasonogram (POCUS) has emerged as a promising modality for real-time monitoring of DD. It offers a more accessible and feasible approach compared to traditional methods, providing immediate feedback on diaphragmatic movement, and facilitates timely intervention. Ultrasound has been used to assess Diaphragmatic Inspiratory Amplitude (DIA) (the expansion of the diaphragm when breathing). DIA has been shown to decrease in the post-operative period after cardiac surgery, which has been well-correlated with the occurrence of POPCs, however, its predictive value has not yet been studied in a cohort of cardiac surgical patients. Hence, we aim to address this gap by exploring the utility of DIA measured by ultrasonogram as a predictive tool in anticipating the occurrence of POPCs. We hypothesize that DIA can predict the occurrence of POPC in cardiac surgical patients. We will recruit 130 patients at University Hospital, London Health Science Centre, to this prospective, observational study.

DETAILED DESCRIPTION:
Cardiac surgery represents a critical intervention for various cardiovascular pathologies, yet it is frequently accompanied by a spectrum of postoperative complications.1 Amongst various morbidities, Post-Operative Pulmonary Complications (POPC) represent a significant clinical challenge leading to adverse outcomes like increased morbidity, mortality, and raised healthcare expenditures.2

Despite significant advancements in surgical methods and perioperative care protocols, POPCs still occur with the reported incidence of 3-16% after Coronary artery bypass grafting and 5-7% after valvular heart surgery.3 POPCs encompass various problems such as atelectasis, pneumonia, cardiogenic pulmonary oedema, acute respiratory distress syndrome, pneumothorax, pleural effusion, phrenic nerve injury and prolonged mechanical ventilation (PMV).2

The diaphragm, as the principal respiratory muscle, plays a pivotal role in maintaining pulmonary function.4 A normal diaphragmatic function is needed for optimal lung re- expansion post cardiac surgery, especially where the work of breathing is high (due to pain etc). Its function is also crucial in aiding efficacious respiratory secretion clearance through adequate coughing.2 Interventions that amplify the inspiratory muscle strength preoperatively (via an incentive spirometer), and usage of Non-invasive ventilation (NIV) in the postoperative period (via mechanical unloading) have demonstrated efficacy in attenuating the incidence of POPCs.2

Diaphragmatic dysfunction (DD) in the perioperative period of Cardiac surgery has an incidence of up to 20%.5 Diaphragmatic dysfunction after cardiac surgery constitutes a complex phenomenon with multifactorial aetiology, encompassing phrenic nerve injury (due to topical ice-slush usage, surgical trauma, or ligation of its blood supply during internal mammary artery dissection) and the deleterious inflammatory sequelae (from high level of cytokines and mitochondrial oxidative stress) associated with cardiopulmonary bypass (CPB).6

Transient diaphragm impairment is a frequent occurrence in the immediate aftermath of cardiac surgery and can be attributed to various perioperative factors, including sternotomy-associated pain, mechanical constraints on thoracic dynamics, electrolyte derangements, and intrathoracic fluid accumulations.7 However, a subset of patients manifest significant DD, which poses distinct challenges in clinical management and may exert profound ramifications on overall outcomes. Understanding the impact of DD on postoperative pulmonary function is imperative for optimizing patient care and clinical outcomes. Its occurrence has been linked to a spectrum of respiratory complications, ranging from pneumonia to difficulty in weaning from mechanical ventilation.7 Despite its clinical significance, it remains an under evaluated cause of POPCs.4

Conventional diagnostic modalities to study DD, notably transdiaphragmatic pressure measurements, furnish valuable insights into diaphragmatic function, albeit encumbered by inherent invasiveness and limitations in discerning unilateral dysfunction.8 In recent years, the advent of point-of-care ultrasonogram (POCUS) has emerged as a promising modality for real-time monitoring of DD. It offers a more accessible and feasible approach compared to traditional methods, providing immediate feedback on diaphragmatic movement, and facilitates timely interventions (like draining a pleural effusion or instituting NIV as needed).9

Ultrasound guided diaphragmatic function has so far been studied through metrics of Diaphragmatic Inspiratory Amplitude (DIA) {also known as diaphragmatic excursion (DE)}and Diaphragmatic thickening/thickening fraction.9 Both the measurements have been shown to decrease in the post operative period of cardiac surgery and are well correlated with occurrence of POPCs.6

The thickening fraction has also been examined for its predictive value and its reliability (in comparison to conventional diagnostic modalities). It has been established as a reliable tool.2 However, it has been observed that the reproducibility, ease of doing it bedside are inferior as compared to DE/DIA with higher interobserver variability plaguing its widespread usage.9 DIA/DE is proven to be an easier measurement in a point of care situation.9 However, its predictive value has so far not been studied in cardiac surgical patient cohort.

Hence, we aim to address this gap by exploring the utility of DIA measured by ultrasonogram as a predictive tool in anticipating the occurrence of POPCs. We hypothesize that DIA can predict the occurrence of POPC in cardiac surgical patients.

Ultrasonographic measurements will be done preoperatively a day before surgery (T0) and on Postoperative day 1(T1) in Cardiac Surgery Recovery Unit (CSRU). Measurements will be done on both right and left sides during Quiet (Q) and Deep (D) breathing in semi- recumbent posture (30-450 recline of the bed).

Three measurements will be taken during both quiet and deep breathing and an average value will be derived (Qavg and Davg). this will be done for both right and left hemidiaphragms (both pre-surgery and post-surgery). So, for each patient a total of 8 diaphragmatic measurements will be obtained (4 in the pre-surgery period and another 4 in post-surgery period).

Measurement technique and definition of Diaphragmatic Inspiratory Amplitude:

All examinations will be performed by Sonosite SII ultrasound machine (FUJIFILM Sonosite Inc, Bothell, WA, USA) using a 3.5- to5 MHz phased array probe or a 3-12 MHz linear probe. The investigator will stand on the right side of the patient. In each patient, to ensure that all measurements are made from the same acoustic window, the distance between probe placement and the lower extremity of the ribcage on the mid-axillary line will be measured and used as the reference site for the subsequent exam in the postoperative period.

Right hemidiaphragm assessment:

The ultrasound probe will be placed on the right anterior chest wall between midclavicular line and anterior axillary line at the ninth intercostal space. The probe will be positioned craniocaudally and will be directed cephalad, medially, and dorsally. This probe orientation and manoeuvring will help visualize the posterior third of hemi-diaphragm (where diaphragmatic movement will be the greatest) in the anterior subcostal view. The diaphragm will be imaged using Brightness mode (B mode). The probe will be adjusted to obtain a continuous trace of the diaphragm against the acoustic window of the liver (with the confluence of the portal vein in view). Once the diaphragm movement is obtained, the settings will be changed to Motion mode (M mode). The cursor in M mode will be placed perpendicular to the diaphragm movement. The sweep speed will be set at 10/second during this examination. The sine wave obtained from diaphragmatic to and from movement will be frozen. The distance from the sine wave's trough to the highest echogenic line and the sine wave's peak to the highest echogenic line will be measured. The DIA value will be obtained as difference between the above two distances. Brightness mode imaging will be repeated after this, with patient taking a deep breath. If the rib shadows interfere with the imaging, the probe will be moved caudally until a good diaphragmatic excursion is possible to image. At that point the measurements will be repeated in M mode during deep breathing.

Left hemidiaphragm measurement:

The probe will be placed on the lateral chest wall on the left side between the anterior and posterior axillary lines. The probe will be positioned in a craniocaudal orientation with a cephalad, medial and dorsal direction. Brightness mode and Motion mode imaging will be performed as described above. DIA measurements will be calculated as elaborated previously.

Patient will be accompanied into the OR once all the consents (anesthesia and surgical) are obtained. Patient will be connected to various monitoring equipment as per American Society of Anesthesiologist's guidelines. All the required invasive cannulae (venous and arterial) will be accessed and secured as per standard institutional protocols. General anaesthesia (GA) will be induced as per Institutional protocols using 2- 5µg/kg of Fentanyl, 20-30µg/kg of midazolam and 2-2.5mg/kg of Propofol for a target Bi- Spectral Index (BIS) of < 60. Muscle relaxation will be obtained using 0.1mg/kg of vecuronium. All patients will receive controlled ventilation with a 6ml/kg tidal volume and positive end expiratory pressure of 5cm water. GA will be maintained with sevoflurane delivered in air+oxygen mixture with a target end-tidal minimum alveolar concentration 0.8-1 and BIS between 40-60. The neuromuscular block will be maintained with intermittent doses of 0.25mg/kg vecuronium guided by neuromuscular monitoring. This is all standard of care.

For all surgeries requiring cardiopulmonary bypass (CPB), the institution and weaning from CPB will be as per standard institutional protocols. Post completion of Surgery, all patients will be shifted to Cardiac Surgical Recovery Unit (CSRU), for further monitoring and management.

Post surgery DIA measurement:

Ultrasound examination will be performed on extubated patients, breathing spontaneously in semi-recumbent posture (30-450 of incline). The measurements will be taken only if patient's pain score on Visual Analog Scale is < 3. If the score is > 3, then patients will be given 15mg/kg paracetamol intravenously and re-assessed 30 minutes later. All patients will be mobilized by second postoperative day.

The general post cardiac surgical care, (like hemodynamic management, decisions of when to extubate, when to institute Non-invasive ventilation (NIV), when to re-intubate, when to provide oxygen therapy) in CSRU will be delivered by the in-charge staff cardiovascular anaesthesiologist and the cardiac anaesthesia fellows who aren't aware of DIA values. The postop pain will be managed using multimodal analgesia approach as per institutional protocol and will be standard of care.

Values that are not obtained on any day due to difficulties with visualization will be considered as missing values. If the values are not obtained for longer than a day for any patient, either due to technical difficulties or the requirement of continuous mechanical ventilatory support beyond the first 48 hours post-surgery, then they were excluded from further analysis. Patients in whom intermittent non-invasive ventilation is required, the values will be obtained when they are off NIV and comfortable. If the patient is receiving continuous NIV throughout the day, then USG will not be done on that day. However, it will be done the next day when patent is off NIV.

POPC will be diagnosed based on European perioperative clinical outcome guidelines10 and they will be graded for their severity based on the Clavien-Dindo11 classification. The three main components of POPC, which are of interest to our study are the occurrence of pneumonia, clinically significant atelectasis, or prolonged mechanical ventilation. These are of particular interest because they have a significant impact on patient outcomes and very possibly are influenced by respiratory muscle strength. Patients will be followed up for the development of POPC till postop day 5 (this includes days in CSRU plus the days in the post cardiac surgical ward) or the day of discharge from hospital (whichever is earlier). POPC diagnosis and assessment will be done by an independent investigator who will not know the DIA values. Observation of patients in this patient population for POPCs following surgery is standard of care.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged>18 years and undergoing elective cardiac surgery.

Exclusion Criteria:

1. . Redo Cardiac surgery.
2. . Pre-existing CNS disease (like Parkinson's disease) or Brain injury or Psychiatric disorder
3. . Emergency cardiac surgery
4. . Surgeries done via Thoracotomy approach.
5. . Pre-surgery ICU stay/ on NIV/ on mechanical ventilation.
6. . Pre-surgery Hemodynamic instability requiring vasopressors/IABP institution.
7. . Age<18
8. . Elevated hemidiaphragm before surgery on chest x ray
9. . Pre-existing neuromuscular disorders (like myasthenia gravis etc.)
10. . Patients planned for heart transplantation.
11. . Patients on mechanical circulatory support preoperatively (intra-aortic balloon pump, extracorporeal membrane oxygenation, or ventricular assist device).
12. . Inability to give consent.

Ages: 19 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients over the age of 18 who present to hospital for elective cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Determine the utility of diagnostic inspiratory amplitude (DIA) as a prognosticator for postoperative pulmonary complications (POPCs). | One day prior to surgery to one day following surgery
  Ultrasonography will be used to measure DIA of patients one day before cardiac surgery and one day after to detect any changes in DIA that occurred and to determine if these changes are associated with POPCs. Occurrence of POPCs will be evaluated by obtaining this data from patient observation.

CONTACTS AND LOCATIONS:
Overall Officials: Raffael Zamper, MD, Principal Investigator — Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moury PH, Cuisinier A, Durand M, Bosson JL, Chavanon O, Payen JF, Jaber S, Albaladejo P. Diaphragm thickening in cardiac surgery: a perioperative prospective ultrasound study. Ann Intensive Care. 2019 Apr 24;9(1):50. doi: 10.1186/s13613-019-0521-z. PMID 31016412
- [Background] Cavayas YA, Eljaiek R, Rodrigue E, Lamarche Y, Girard M, Wang HT, Levesque S, Denault AY. Preoperative Diaphragm Function Is Associated With Postoperative Pulmonary Complications After Cardiac Surgery. Crit Care Med. 2019 Dec;47(12):e966-e974. doi: 10.1097/CCM.0000000000004027. PMID 31609771
- [Background] Naveed A, Azam H, Murtaza HG, Ahmad RA, Baig MAR. Incidence and risk factors of Pulmonary Complications after Cardiopulmonary bypass. Pak J Med Sci. 2017 Jul-Aug;33(4):993-996. doi: 10.12669/pjms.334.12846. PMID 29067080
- [Background] Vanamail PV, Balakrishnan K, Prahlad S, Chockalingam P, Dash R, Soundararajan DK. Ultrasonographic Assessment of Diaphragmatic Inspiratory Amplitude and Its Association with Postoperative Pulmonary Complications in Upper Abdominal Surgery: A Prospective, Longitudinal, Observational Study. Indian J Crit Care Med. 2021 Sep;25(9):1031-1039. doi: 10.5005/jp-journals-10071-23962. PMID 34963722
- [Background] Pasero D, Costamagna A, Marchisio A, Pivetta E, Giunta M, Fanelli V, Brazzi L. Diaphragmatic dysfunction following cardiac surgery: Observational study. Eur J Anaesthesiol. 2019 Aug;36(8):612-613. doi: 10.1097/EJA.0000000000000969. No abstract available. PMID 31274546
- [Background] Bruni A, Garofalo E, Pasin L, Serraino GF, Cammarota G, Longhini F, Landoni G, Lembo R, Mastroroberto P, Navalesi P; MaGIC (Magna Graecia Intensive care and Cardiac surgery) Group. Diaphragmatic Dysfunction After Elective Cardiac Surgery: A Prospective Observational Study. J Cardiothorac Vasc Anesth. 2020 Dec;34(12):3336-3344. doi: 10.1053/j.jvca.2020.06.038. Epub 2020 Jun 17. PMID 32653270
- [Background] Laghlam D, Naudin C, Srour A, Monsonego R, Malvy J, Rahoual G, Squara P, Nguyen LS, Estagnasie P. Persistent diaphragm dysfunction after cardiac surgery is associated with adverse respiratory outcomes: a prospective observational ultrasound study. Can J Anaesth. 2023 Feb;70(2):228-236. doi: 10.1007/s12630-022-02360-8. Epub 2022 Dec 13. PMID 36513852
- [Background] Lerolle N, Guerot E, Dimassi S, Zegdi R, Faisy C, Fagon JY, Diehl JL. Ultrasonographic diagnostic criterion for severe diaphragmatic dysfunction after cardiac surgery. Chest. 2009 Feb;135(2):401-407. doi: 10.1378/chest.08-1531. Epub 2008 Aug 27. PMID 18753469
- [Background] Tralhao A, Cavaleiro P, Arrigo M, Lopes JP, Lebrun M, Rivas-Lasarte M, Le Pimpec-Barthes F, Latremouille C, Achouh P, Pirracchio R, Cholley B. Early changes in diaphragmatic function evaluated using ultrasound in cardiac surgery patients: a cohort study. J Clin Monit Comput. 2020 Jun;34(3):559-566. doi: 10.1007/s10877-019-00350-8. Epub 2019 Jul 5. PMID 31278543
- [Background] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542